CLINICAL TRIAL: NCT03705065
Title: A Phase 4, Randomized, Open-Label Study of the Pharmacokinetics and Tolerability of Bupivacaine HCl Following One of Two Routes of Administration in Subjects Undergoing Augmentation Mammoplasty
Brief Title: Bupivacaine HCl PK and Safety in Augmentation Mammoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUPI-502
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Analgesia
Keywords: augmentation mammoplasty
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1 (Experimental): Bupivacaine HCI by instillation into each pectoral pocket.
  Interventions: Drug: Bupivacaine HCl
- Treatment Group 2 (Experimental): Bupivacaine HCI by injection into each pectoral pocket.
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: Bupivacaine HCl — Bupivacaine HCl without epinephrine 0.25%, 60 mL (30 mL per pectoral pocket)

SUMMARY:
This is a Phase 4, randomized, open-label study of bupivacaine HCl administered either by instillation into the surgical site or by injection into the surgical site in subjects undergoing bilateral submuscular augmentation mammoplasty under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo primary bilateral submuscular augmentation mammoplasty with saline or silicone smooth implants with a volume of 300 to 500 mL, inclusive.
* Has an American Society of Anesthesiologists Physical Status of I, II, or III.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Has a planned concurrent surgical procedure (eg, mastopexy).
* Has a planned concurrent reconstructive procedure status post breast cancer therapy.
* Has a pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain that is not strictly related to the augmentation mammoplasty.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has been administered any local anesthetic within 72 hours prior to the scheduled surgery.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* As per subject history and/or medical records, has active infection or is currently undergoing treatment for Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV).
* Has uncontrolled anxiety, psychiatric, or neurological disorder.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention-deficit/hyperactivity disorder, benzodiazepine for anxiety disorder) may be eligible for participation in the study at the discretion of the Sponsor. Subjects taking any marijuana (medical or recreational) are not allowed to participate in the study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half-lives.
* Has undergone 3 or more surgeries within 12 months.
* Has a body mass index (BMI) >35 kg/m2.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Baseline through 72 hours after start of study drug administration
Area Under the Concentration-time Curve From Time 0 to the Last Collection Time After Study Drug Administration (AUC Last) | Baseline through 72 hours after start of study drug administration
Area Under the Concentration-time Curve From Time 0 to Infinity After Study Drug Administration (AUC∞) | Baseline through 72 hours after start of study drug administration
Time to Maximum Plasma Concentration (Tmax) | Baseline through 72 hours after start of study drug administration
The Apparent Terminal Elimination Rate Constant (λz) | Baseline through 72 hours after start of study drug administration
The Apparent Terminal Elimination Half-life (t1/2el) | Baseline through 72 hours after start of study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Hermann Drive Surgical Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided